CLINICAL TRIAL: NCT00082602
Title: Galantamine ER Open Label Rapid Dose Escalation Trial in Alzheimer's Disease
Brief Title: Safety and Tolerability Study of Extended Release (ER) Galantamine in Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004699
Record Dates: First submitted 2004-05-12; First posted 2004-05-17 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2009-04

CONDITIONS: Alzheimer's Disease
Keywords: galantamine; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: galantamine ER

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of an extended release formulation of the drug galantamine using a rapid dose escalation regimen.

DETAILED DESCRIPTION:
To improve dosing convenience of the current formulation of galantamine, a new once daily dosing Extended Release (ER) formulation was developed. In a different large study, in which approximately 900 patients with Alzheimer's disease participated, efficacy of the Extended Release formulation was confirmed. During the first 8 weeks of treatment, nausea and vomiting occurred less frequently with the Extended Release than Intermittent Release formulation. This suggests that patients might better tolerate a rapid dose escalation to the initial maintenance dose of 16mg daily, thereby improving the risk/benefit ratio during the first 4 weeks of therapy, i.e. receiving more drug sooner. The trial objectives are: 1) to demonstrate the safety and tolerability of galantamine Extended Release 16 mg daily when titrated from 8 mg daily after one week; 2) to evaluate the effect of galantamine Extended Release on cognition as measured by the Mini Mental State Examination. Results from prior trials show that galantamine Intermittent Release (twice a day dosing) has a high rate of adverse events when dose escalations occur at one-week intervals. Therefore, current galantamine labelling recommends that the drug dose be escalated once every 4 weeks. The study hypotheis is that the rapid dose escalation of the Extended Release formulation in subjects with Alzheimer's disease is safe and well tolerated. Comparison of adverse event rates will be made to the first 8 weeks Reminyl Extended Release group of another trial in which the Extended Release formulation was titrated from 8 mg daily to 16 mg daily at 4 weeks. Subjects will receive galantamine Extended Release capsules by mouth starting at 8 mg daily and after one week will be titrated up to 16 mg daily. This dose will be maintained for 11 additional weeks.

8 mg of Galantamine Extended Release Capsules once daily for one week. After one week will be titrated up to 16 mg daily for 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients diagnosed with Alzheimer's Disease
* Age >= 60 years
* Presence of mild to moderate dementia as evidenced by Mini Mental State Examination (MMSE) score of 10-24 inclusive at screening
* History of cognitive decline that had been gradual in onset and progressive over a period of at least six months

Exclusion Criteria:

* Neurodegenerative disorders
* One of the following conditions possibly resulting in cognitive impairment: Acute cerebral trauma or injuries secondary to chronic trauma (such as boxing), hypoxic cerebral damage, whether or not due to acute or chronic cerebral hypoperfusion
* Vitamin deficiency states, such as folate, vitamin B12 or other B complex deficiencies
* Neurosyphilis or other infections resulting in cerebral abscesses, meningitis, or encephalitides such as AIDS
* Primary or metastatic cerebral neoplasia
* Significant endocrine or metabolic disease e.g., untreated or uncontrolled thyroid, parathyroid or pituitary disease, Cushing's syndrome, severe renal failure or uncontrolled diabetes mellitus
* Mental retardation or oligophrenia
* Multi-infarct dementia or clinically active cerebrovascular disease as evidenced by: a history of a significant cerebrovascular event yielding a physical or neurologic deficit likely to confound the assessment of the subject's intellectual function, multiple focal signs on neurological examination indicative of multiple ischemic attacks, significant findings on an available CT or MRI scan taken within the last 12 months
* Subjects with the following co-existing medical conditions: Any history of epilepsy or convulsions except for febrile convulsions during childhood
* Current clinically significant psychiatric disease, in particular current major depression, schizophrenia, bipolar disorder, moderate to severe or uncontrolled behavioral disturbances
* Peptic ulcer disease: if the ulcer is considered to be still active, or if treatment is not successful (symptoms present)
* Clinically significant hepatic, renal, pulmonary, metabolic or endocrine disturbances
* Clinically significant urinary outflow obstruction
* Current, clinically significant cardiovascular disease that would be expected to limit the subject's ability to participate in and complete a 12-Week trial. The following would usually be considered clinically significant cardiovascular diseases: cardiac surgery or myocardial infarction within the past 6 months, angina or coronary artery disease that required a change in anti-angina medication within the last 3 months, decompensated congestive heart failure, cardiac disease potentially resulting in syncope, near syncope or other alterations of mental status, atrial fibrillation, bradycardia < 50/min., atrio-ventricular block > first degree
* Severe mitral or aortic valvular disease
* Uncontrolled high blood pressure (systolic blood pressure > 170 mmHg or diastolic blood pressure > 110 mmHg) or sustained hypotension
* Any agent being used for the treatment of dementia (approved, experimental or over the counter agents
* Subjects who have previously received Cognexâ, Ariceptâ, metrifonate, Exelonâ, Reminyl, or Namendaâ for treatment of Alzheimer's disease, no matter if approved or experimental can be included in this trial provided that during the 30 days prior to baseline they were not taking these agents
* O History of drug or alcohol abuse within the last year or prior prolonged history of the same
* Female subjects of childbearing potential
* Subjects who in the opinion of the investigator are otherwise unsuitable for a trial of this type
* History of severe drug allergy or hypersensitivity, including recorded hypersensitivity to cholinesterase inhibitors, choline agonists or identical agents, or bromide
* Subjects who have previously been enrolled in other galantamine trials
* Subjects who have received an investigational medication within the last 30 days
* Conditions that could interfere with the absorption of the compound or with the evaluation of the disease
* Employees of the investigator

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2004-05; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
The primary end point occurs at Week 8. The primary outcome measures will be tolerability and safety through rates of adverse events.

SECONDARY OUTCOMES:
The secondary end point occurs at Week 12. The secondary outcome measure will be the Mini Mental State Examination score.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Safety and Tolerability Study of Extended Release (ER) Galantamine in Alzheimer's Disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=625&filename=CR004699_CSR.pdf